CLINICAL TRIAL: NCT03239457
Title: Efficacy and Safety of Heberprot-P® in Patients With Advanced Diabetic Foot Ulcer in Dasman Diabetes Institute. Demonstrative Study
Brief Title: Efficacy and Safety of Heberprot-P® in Patients With Advanced Diabetic Foot Ulcer in Dasman Diabetes Institute.
Status: Completed | Type: Observational
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: Cuban Center for Genetic Engineering and Biotechnology (Other)
Responsible Party: Sponsor
Other Study IDs: RA 2014-051
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2016-05

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Heberprot P treatment: Patients with diabetic foot ulcers treated with Heberprot P
  Interventions: Biological: Heberprot P

INTERVENTIONS:
Biological: Heberprot P — 75 µg vials administered at the rate of a vial 3 times per week (Sunday Tuesday, Thursday) by intralesional and perilesional route.For this, the reconstitution and dilution of the vial will be carried out with 5 mL of water for injection. The administrations will be kept up to 8 weeks of treatment or until there is achieved granulation of the 100 % of the lesion.
  Other Names: Human recombinant Epidermal Growth Factor

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the intralesional administration of Heberprot-P® (human recombinant epidermal growth factor) plus the standard treatment in patients with complex diabetic foot and risk of major amputation in Kuwait.

DETAILED DESCRIPTION:
Diabetic foot ulcers constitute an important medical problem in the patients with diabetes mellitus. The epidermal growth factor (EGF) stimulates the proliferation of fibroblasts, keratinocytes and vessel endothelial cells, which contributes to its healing properties.In previous phase I-III clinical studies in patients with diabetic foot ulcers grade 3 and 4 of the Wagner's classification (Meggitt-Wagner classification), it has been demonstrated that the intralesional administration of the EGF stimulates the healing, having as result the formation of a useful granulation tissue in the bed of the ulcers and the later closure of the lesion. This effect was associated with a decreased risk of amputation. Considering the pharmacological actions identified for the EGF, the pathogenesis of the disease, previous clinical results and the absence of an effective treatment for this condition justifies the current clinical study. The purpose of this study is to assess the efficacy and safety of the intralesional administration of Heberprot-P® (human recombinant epidermal growth factor) plus the standard treatment in patients with complex diabetic foot and risk of major amputation in Kuwait.

A demonstrative study, open, single-center, uncontrolled, with one treatment group to be conducted in a maximum of 50 patients with DFU. The study will be conducted at DDI, Kuwait.

General objective To assess the efficacy and safety of the intralesional administration of Heberprot-P® plus the standard treatment in patients with diabetic foot ulcer in University of Texas Wound Classification AI-AII and CI-CII and risk of major amputation.

Specific objectives To determine the efficacy of Heberprot-P® in patients with diabetic foot ulcer in terms of the proportion of patients that reach complete response (100% of the area covered by granulation tissue) at the end of treatment.

To determine the time to reach the granulation tissue 100% of the lesion area. To assess the effect of the administration of Heberprot-P® in the prevention of major amputations.

To identify and characterize the adverse events associated with the intralesional and perilesional administration of Heberprot-P® in patients with diabetic foot.

Methods to evaluate the quality of the assessment procedures of the efficacy. Quality control visits will be carried out during the demonstration by the Research affairs office in DDI, Kuwait and CIGB, previously coordinated with the investigators. When the patient finishes the treatment, the monitors will gather the CRFs leaving a copy in the research site.

Behavior in case of exit from the demonstration Management of withdrawals and missings to evaluation visits is explained in item. The assessment will be carried out according to the principle of intent to treat, so all the patients once included will be considered in the response assessment, regardless they have had received the treatment or not, or having completed the follow-up.

Adverse events to that can appear and their recording An adverse event is any medical undesirable and not deliberate manifestation that happens in a patient or subject of a clinical research to which a drug has been administered, regardless if it is related or not to this treatment.

This way, it can be any sign (including for example abnormal laboratory data), symptoms or disease associated temporarily with the use of a pharmaceutical product, being or not a causality ratio. The exacerbations of symptoms/diseases that were present before the study will also be included as adverse events.

In the post-marketing stage, during the active pharmaco-surveillance of the use of Heberprot-P® there were included about 4000 subjects. In the initial analysis of 1851 patients, 873 patients reported adverse events, the most frequent were: pain at the site of application (21.7%), shivering from cold (19.8), burning at the application site (16.0%), chills (9.2%), local infection (3.8%) and fever (2.3%).

All the information related to the occurrence of adverse events presented in the patients included in the clinical demonstration will be registered and described by the researchers in the Adverse Events Form of the CRF. There will be described the type, duration, intensity, seriousness, causality and the followed behavior.

The intensity (severity) will be classified the following way:

1. Mild: adverse event that the subject tolerates well, causes minimal inconveniences and does not interfere with the daily activities.It does not need treatment and does not interrupt the administration.
2. Moderate: adverse event that is annoying enough as to interfere the daily activities. It needs treatment and not necessarily needs the suspension of the causative drug.
3. Severe: adverse event that prevents from doing the daily activities.

The criteria that will be used to define an adverse event as serious will include the presence of some of the following conditions:

It endangers the subject's life causes the death causes or prolongs the hospitalization produces disability/incapacity causes congenital anomaly

These events need the suspension of the causative drug.

Behavior in case of adverse events The most frequent clinical adverse events reported with the use of Heberprot-P are pain and Burning sensation in the injection site, shivering, chills, local infection and fever. The behavior in case of these adverse events includes the administration of antibiotics.

In case allergic reactions appear, the behavior will depend on their magnitude, including the use of antihistamines, steroids or even definitive suspension of the treatment.

In case of having serious adverse events, the treatment will be suspended, there will be taken the measures needed depending on the type of event and it will be considered the possible expeditious report of the event.

Expeditious report of the adverse events Any unexpected serious adverse event that appears in the course of the clinical demonstration will be valued with a view to the expeditious report. The term "unexpected" refers to the events which specificity or seriousness is not consistent with the available information of the product (Annex 3).

In case you have a serious and unexpected adverse effect, the Clinical investigator will report to Dr Rafael Ibargollin Ulloa and DDI Ethics committee .

Follow up as for all reportable AEs. Basic follow up information must also be documented on the SAE Report Form and in the CRF.

Recording of the information and handling the data

* Researcher´s registry. After the patient has been included Patient´s identification data.
* Registry of Included and Not included Patients. During the whole period of inclusion of cases List of all the patients with diagnosis who come to the participant service, indicating if they were included or not and the causes of non-inclusion.
* Informed consent Before the inclusion Record of the patient's voluntariness in taking part in the study.
* Case Report Form. At the beginning and during the patient's follow-up. General data, clinical assessments and complementary examinations.
* Serious adverse event notification form. When serious and unexpected adverse events are faced. Patient's data, description of the adverse events, date and time of start and completion, behavior, causality ratio and result.

The information specified in the CRF will be completed by researchers in each of the assessments. When patients have completed follow-up, the CRF should be reviewed and signed. The CRF will be filled in duplicate, the researcher will keep a copy and send the other to the monitors in the CIGB. Informed consent will also fill in duplicate, one for the investigator and the other to the patient.

With the individual data a database will be created, which will serve for their processing. A double entry of the data will be carried out for later comparison and correction from possible errors.

Procedure for preserving the information The CRFs, the databases, the reports that are generated and the compact discs with the images will be preserved in the site destined for this effect, previously designated by the persons in charge of the demonstration and they will be preserved for at least 15 years by the sponsor.

Exploratory analysis of the data The analyses will be carried out by intention to treat, considering the abandonments as non-responses to the treatment.

With each variable (main, secondary and control) exploratory analyses will be carried out to know their global behavior and to evaluate fulfillment of the necessary hypothesis in order to apply the proper statistical tests in the assessment stage.With the quantitative variables, the assumptions of homogeneity of variances (Levene's test) and of approximation to a normal distribution (Shapiro-Wilk's test) must be verified. Additionally, as measurements of central tendency and dispersion, the mean, median, standard deviation, interquartile range and minimum and maximum values will be estimated. With the qualitative variables, the distribution of frequencies should be estimated. It is proposed to carry out a Cluster Analysis as exploratory method of association between the variables.

Homogeneity of the sample With the qualitative variables (sex, type of Diabetes Mellitus, obesity, smoking arterial hypertension, structural deformities, consumption of alcohol, current treatment for the diabetes, history of ulcers, location of the lesion, osteomyelitis, DDI, University of Texas Wound Classification System.

The frequency distribution will be estimated. With the quantitative variables (age, time of evolution of the diabetes mellitus and of the ulcer, glycosylated hemoglobin, initial area of the lesion, ankle/arm pressure index at the beginning): The measurements of central tendency and dispersion will be estimated and analysis of normality will by made (Shapiro-Wilk's tries) and of homogeneity of variances (Levene's test).

With all (quantitative and qualitative variables): A logistic regression model will be adjusted to study the influence of each of them and their interactions on the response to the treatment and occurrence of serious adverse events. In case any statistically significant dependence(s) is/are detected, the confirmatory analysis with the main variable should envisage it/them as covariable (s) or stratum (strata).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of diabetic foot ulcer,University of Texas Wound Classification AI-AII and CI-CII with or without ischemia at least of 4 weeks of evolution Ulcers with an area between ≥ 2 cm2 or greater (after sharp debridement of free, non-viable, hyperkeratotic and fibrotic tissue) Patients with age than 22 years. Voluntariness of the patient by signing up the informed consent, and written form signed the date prior to study.

Exclusion Criteria:

Hemoglobin ≤100 g/L. Patients with a significant acute cardiovascular event (Major Acute Cardiovascular Event) within 3 months prior such as acute myocardial infarction, severe angina pectoris, acute stroke or transient ischemic attack, and/or thrombo-embolism event.

Patients with chronic uncompensated diseases: diabetic coma, or renal failure (creatinine 200 mmol/L and oligoanuria).

Antecedents or suspicion of malignant diseases (general physical examination, rectal tact, examination of breast, abdominal ultrasound, thorax radiography and blood hemochemistry).

Psychiatric diseases that compromise the treatment or the evaluations Infection Pregnancy or breastfeeding.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of the State of Kuwait attending to Dasman Diabetes Institute with Diabetic foot ulcer (DFU)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with 100% of the lesion area covered by granulation tissue. | The total duration of patient participation in the study will be 8 weeks for intervention or earlier if they show 100% granulation. Patients will be followed up until 20 weeks for final assessment
  Lesion area granulation will be assessed as: Non response (0%-25%); Minimal (25%-50%); Partial (50%-75%); Total (75%-100%)

SECONDARY OUTCOMES:
Time in which the formation of the granulation tissue 100% | 8 weeks
Need of major amputation | 20 weeks
Adverse events | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ibargollín Ulloa, MD, MSc, Principal Investigator — Cuban Center for Genetic Engineering and Biotechnology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Boulton AJ, Kirsner RS, Vileikyte L. Clinical practice. Neuropathic diabetic foot ulcers. N Engl J Med. 2004 Jul 1;351(1):48-55. doi: 10.1056/NEJMcp032966. No abstract available. PMID 15229307
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Reiber GE. The epidemiology of diabetic foot problems. Diabet Med. 1996;13 Suppl 1:S6-11. No abstract available. PMID 8741821
- [Background] Lipsky BA. Medical treatment of diabetic foot infections. Clin Infect Dis. 2004 Aug 1;39 Suppl 2:S104-14. doi: 10.1086/383271. PMID 15306988
- [Background] Dinh TL, Veves A. A review of the mechanisms implicated in the pathogenesis of the diabetic foot. Int J Low Extrem Wounds. 2005 Sep;4(3):154-9. doi: 10.1177/1534734605280130. PMID 16100096
- [Background] Simmons Z, Feldman EL. Update on diabetic neuropathy. Curr Opin Neurol. 2002 Oct;15(5):595-603. doi: 10.1097/00019052-200210000-00010. PMID 12352003
- [Background] Reiber GE, Vileikyte L, Boyko EJ, del Aguila M, Smith DG, Lavery LA, Boulton AJ. Causal pathways for incident lower-extremity ulcers in patients with diabetes from two settings. Diabetes Care. 1999 Jan;22(1):157-62. doi: 10.2337/diacare.22.1.157. PMID 10333919
- [Background] Lavery LA, Armstrong DG, Murdoch DP, Peters EJ, Lipsky BA. Validation of the Infectious Diseases Society of America's diabetic foot infection classification system. Clin Infect Dis. 2007 Feb 15;44(4):562-5. doi: 10.1086/511036. Epub 2007 Jan 17. PMID 17243061
- [Background] Brem H, Sheehan P, Boulton AJ. Protocol for treatment of diabetic foot ulcers. Am J Surg. 2004 May;187(5A):1S-10S. doi: 10.1016/S0002-9610(03)00299-X. PMID 15147985
- [Background] Williams DT, Hilton JR, Harding KG. Diagnosing foot infection in diabetes. Clin Infect Dis. 2004 Aug 1;39 Suppl 2:S83-6. doi: 10.1086/383267. PMID 15306984
- [Background] Eldor R, Raz I, Ben Yehuda A, Boulton AJ. New and experimental approaches to treatment of diabetic foot ulcers: a comprehensive review of emerging treatment strategies. Diabet Med. 2004 Nov;21(11):1161-73. doi: 10.1111/j.1464-5491.2004.01358.x. PMID 15498081
- [Background] COHEN S. Isolation of a mouse submaxillary gland protein accelerating incisor eruption and eyelid opening in the new-born animal. J Biol Chem. 1962 May;237:1555-62. No abstract available. PMID 13880319
- [Background] Cohen S, Carpenter G. Human epidermal growth factor: isolation and chemical and biological properties. Proc Natl Acad Sci U S A. 1975 Apr;72(4):1317-21. doi: 10.1073/pnas.72.4.1317. PMID 1055407
- [Background] Cohen S, Carpenter G, King L Jr. Epidermal growth factor-receptor-protein kinase interactions. Prog Clin Biol Res. 1981;66 Pt A:557-67. PMID 6273929
- [Background] Gospodarowicz D. Epidermal and nerve growth factors in mammalian development. Annu Rev Physiol. 1981;43:251-63. doi: 10.1146/annurev.ph.43.030181.001343. No abstract available. PMID 7011183
- [Background] Gross I, Dynia DW, Rooney SA, Smart DA, Warshaw JB, Sissom JF, Hoath SB. Influence of epidermal growth factor on fetal rat lung development in vitro. Pediatr Res. 1986 May;20(5):473-7. doi: 10.1203/00006450-198605000-00018. PMID 3487067
- [Background] Brown GL, Curtsinger L 3rd, Brightwell JR, Ackerman DM, Tobin GR, Polk HC Jr, George-Nascimento C, Valenzuela P, Schultz GS. Enhancement of epidermal regeneration by biosynthetic epidermal growth factor. J Exp Med. 1986 May 1;163(5):1319-24. doi: 10.1084/jem.163.5.1319. PMID 3486247
- [Background] Cohen S, Carpenter G, King L Jr. Epidermal growth factor-receptor-protein kinase interactions. Co-purification of receptor and epidermal growth factor-enhanced phosphorylation activity. J Biol Chem. 1980 May 25;255(10):4834-42. PMID 6246084